CLINICAL TRIAL: NCT02302482
Title: Predictive Factors of the Autonomy Level Change Related to Memory Disorders
Brief Title: Predictive Factors and Autonomy Level Change
Acronym: MEMORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014.868
Record Dates: First submitted 2014-11-14; First posted 2014-11-27 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Memory Impairment
Keywords: Alzheimer's disease or related disorders; Functional autonomy level; Cognitive function; Predictive factors
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional autonomy level collection (Experimental): Collection of the Functional autonomy level every 6 - 12 months by phone
  Interventions: Other: The Lawton Instrumental Activities of Daily Living score (IADL), and the disability assessment of dementia score (DAD-6

INTERVENTIONS:
Other: The Lawton Instrumental Activities of Daily Living score (IADL), and the disability assessment of dementia score (DAD-6

SUMMARY:
The Alzheimer's disease or related disorders (ADRD) are among the most disabling diseases because of their main features such as cognitive impairment, loss of functional autonomy and behavioural disorders. In absence of current curative treatment, the identification of the predictive risk factors of progression of the disease, evaluated through its main symptoms, represents a major stake of public health. The investigators aimed at developing a database, which includes the patient medical records on a prospective basis, in collaboration with the medical and administrative personal and with the University hospital computer science department. The main objective is to study the predictive factors associated with the change of functional autonomy level, measured every 6 months to 12 months by phone, in a Memory Clinic. The study population would consist in about 1000 patients with ADRD. The length of follow-up of each patient will be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo a medical visit in the Memory Clinic for the 1st time
* Patients living at home or in housing
* Patients with memory impairment, at all stage of the disease

Exclusion Criteria:

* Patients in institution
* Patients under legal protection
* Patients with a hearing or visual impairment, which dot not allow to carry out the examination

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10860 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Functional autonomy level | 3 years
  The scores of "Lawton Instrumental Activities of Daily Living" (IADL) and of "Disability Assessment of Dementia" (DAD-6)

SECONDARY OUTCOMES:
Cognitive function level | 3 years
  Mini Mental Test examination (MMSE)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Dugoujon, Caluire-et-Cuire
  - Hospices Civils de Lyon - Hôpital des Charpennes, Lyon

REFERENCES:
- [Derived] Dauphinot V, Moutet C, Rouch I, Verdurand M, Mouchoux C, Delphin-Combe F, Gaujard S, Krolak-Salmon P; MEMORA group. A multicenter cohort study to investigate the factors associated with functional autonomy change in patients with cognitive complaint or neurocognitive disorders: the MEMORA study protocol. BMC Geriatr. 2019 Jul 18;19(1):191. doi: 10.1186/s12877-019-1204-1. PMID 31319809